CLINICAL TRIAL: NCT06408402
Title: Impact of Environmental Exposures on Tumor Risk in Subjects at Risk of Hereditary SDHx-related Paragangliomas - National Study
Brief Title: Impact of Environmental Exposures on Tumor Risk in SDHx-mutation Carriers
Acronym: PGLEXPO2
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); ANSES (Other); Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230878; HGT/MFI/AR245071 (Other: Commission Nationale de l'Informatique et des Libertés); 2023-A02297-38 (Other: Agence Nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2024-03-27; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: SDH-Related Familial Paraganglioma; SDHx-Related Syndromes; SDH Gene Mutation; Environmental Exposure
Keywords: hereditary paraganglioma; SDHx gene mutation; environmental exposure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample (10 ml on EDTA) will be proposed to the participants to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases: SDHx mutation carriers diagnosed for a SDHx-related tumor
- Controls: Controls : SDHx mutation carriers with no SDHx-related tumor

SUMMARY:
The primary objective of the PGL.EXPO-2 study is to test the hypothesis that exposure (occupational, environmental and/or domestic) to succinate dehydrogenase inhibitors (SDHi) could contribute to tumor emergence in subjects carrying a germline mutation in one of the SDHx genes.The primary endpoint will be the proportion of subjects (cases or controls) exposed to SDHi and the association with paraganglioma risk.

In addition, a blood sample (10 ml on EDTA) will be proposed to the participants to the study

DETAILED DESCRIPTION:
Patients will be selected from subjects with a mutation in one of the SDHx genes. The cases will have developed a tumor, while the controls will be tumor-free. Controls will be matched to the cases according to age and type of gene affected. Past exposures will be sought through a telephone questionnaire.

In addition, a blood sample (10 ml on EDTA) will be proposed to the participants to the study

ELIGIBILITY:
Inclusion Criteria:

* Cases: SDHx mutation carriers diagnosed for a SDHx-related tumor
* Controls: SDHx mutation carriers with no SDHx-related tumor

Exclusion Criteria:

* Incapacity to exercise free and informed consent for the study
* Patient under tutorship or guardianship or legal safeguard

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 650 cases and 650 controls will be enrolled in different French referral centers where they are regularly managed and followed for a SDHx-related tumor risk. They will be matched on their date of birth
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Impact of SDHi exposure in paraganglioma occurence | 36 months
  Association between exposures and tumor occurrence measure with Odd ratio

SECONDARY OUTCOMES:
Spatial distribution of cases | 48 months
  Spatial distribution of tumor incidence
Incidence rate in France of pathologies linked to SDHx gene mutations | 48 months
  Incidence rate in France of pathologies linked to SDHx gene mutations

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Paule Gimenez-Roqueplo, MD, PhD, Study Director — Hôpital européen Georges Pompidou - APHP
Locations (19):
- France (19):
  - CHU d'Angers, Angers
  - CHU Jean Minjoz Besançon, Besançon
  - Hôpital Louis Pradel, Bron
  - CHU de Caen, Caen
  - Hôpital Michalon - CHU Grenoble, Grenoble
  - CHU de Lille - Hôpital HURIEZ, Lille
  - Hopital de la Conception - Marseille, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice -Hôpital Archet 2, Nice
  - Hôpital Pitié-Salpêtrière - APHP, Paris
  - Hôpital Cochin - APHP, Paris
  - Hôpital européen Georges Pompidou - APHP, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rennes - Hôpital Sud, Rennes
  - Hôpitaux universitaire de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHU de Toulouse - Hôpita Larrey, Toulouse
  - CHU Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).